CLINICAL TRIAL: NCT01430234
Title: Enzyme Substitution in Exocrine Pancreatic Insufficiency; Self Administration Against a Fixed Dose Regimen
Brief Title: Enzyme Suppletion in Exocrine Pancreatic Dysfunction
Acronym: SAPES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Foundation for Liver Research (Other)
Collaborators: Axcan Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SAPES
Record Dates: First submitted 2011-09-01; First posted 2011-09-08 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Pancreatitis; Exocrine Pancreatic Insufficiency
Keywords: Chronic pancreatitis; Exocrine insufficiency; Pancreatic enzyme replacement therapy; Self-administration
MeSH Terms: conditions — Pancreatitis, Chronic; Exocrine Pancreatic Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Panzytrat fixed dose vs. self-dosing (Other): In Phase I (week 1-4) patients will use the fixed amount of lipase as was prescribed by their treating physician. Phase II (week 5-9) patients will start the self-dosage regimen with pancreatic enzymes (without exceeding the maximum amount of 16 capsules per day). They are properly educated by the researcher and dietician how to adjust the amount of pancreatic enzymes to the fat intake in their diet.
  Interventions: Drug: Panzytrat 25.000 FIP-E units of Lipase

INTERVENTIONS:
Drug: Panzytrat 25.000 FIP-E units of Lipase — patients will experiment with Panzytrat (containing 25.000 units of lipase) to a maximum of 16 capsules a day according to general guidelines.
  Other Names: Pancreatine of porcine-origin

SUMMARY:
Treatment of exocrine insufficiency (EPI) consists of pancreatic enzyme replacement according to the fat intake. Prescribing a sufficient dose of pancreatic enzymes is mandatory for the treatment to be effective. In addition, consultation of a specialized dietician is pivotal to educate patients about the proper use of pancreatic enzymes. However, based on a recent prospective survey in the Netherlands amongst chronic pancreatitis patients, it seems that enzymes are underused and a dietician is seldom consulted. The aim of this study is to assess if there is a difference in efficacy of pancreatic enzymes in a self-dosage regimen after extensive patient-education in comparison to the standard treatment for patients with EPI.

DETAILED DESCRIPTION:
This is a prospective, open, comparative study with a linear design with two sequential phases (observatory, then patient-monitored).

The research population consists of patients who are treated with pancreatic enzymes (< 6 capsules p/d containing 25,000 units of lipase) for exocrine insufficiency caused by chronic pancreatitis.

After inclusion, patients will discontinue taking pancreatic enzymes during one week (wash-out period). The last four days of this week, a fecal fat balance test will be performed to quantify the fecal fat loss without enzyme correction. If the fecal fat excretion is less than 15%, this is considered normal and therefore the patient will be excluded from the study. Subsequently, the next three weeks of the trial the patient will restart using the same dose of pancreatic enzymes the way it was prescribed before inclusion. The last four days of the fourth week, a fecal fat balance test will be repeated to quantify the fecal fat loss with enzyme correction. After this test the intervention takes place, consisting of a standardised education of the patient by a dietician. In the second phase of four weeks, patients are stimulated to use this information to self-dose the amount of pancreatic enzymes according to the fat content of their diet. In the last week of the study a fecal fat balance test will be repeated.

The primary endpoint is the fecal fat excretion. Secondary endpoints are the change in enzyme dose after intervention, improvement of complaints (e.g. steatorrhoea related complaints, abdominal cramps, abdominal pain), change in dietary habits, patient satisfaction, quality of life, evaluation of the nutritional status, and the occurrence of side effects.

Because the maximum amount of 16 capsules of pancreatic enzymes a day according to the standard guidelines will not be exceeded in this trial, no risks are foreseen. The anticipated benefit of the study is that patients will be treated more effectively for their EPI. The burden of this trial for patients is the repeated fecal fat balance test.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years.
* EPI caused by CP.
* Treated with enzyme therapy (≤ 6 capsules of 25.000 FIP-E units of lipase per day).
* Fecal elastase < 0.200 mg/g
* fecal fat-absorption < 85% without using enzymes.

Exclusion Criteria:

* Subjects who are unwilling or unable to understand and participate in the study and/or sign the informed consent.
* Any known gastro-intestinal disease or major gastrointestinal or pancreatic surgery that could potentially affect the intestinal absorption or metabolism of fat
* Gastroparesis of any aetiology
* Hypersensitivity to pork protein
* Acute pancreatitis
* Limited life-expectancy of ≤ 6 months
* Malignancy of the pancreas
* Pregnancy/lactation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Fecal Fat percentage | week 1, 5 and 9
  difference in efficacy measured by the fecal fat content during treatment with pancreatic enzymes in a self-dosage regimen after extensive patient-education in comparison to the standard treatment for patients with EPI due to chronic pancreatitis

SECONDARY OUTCOMES:
enzyme dose | On a weekly base during 9 weeks
  Change in enzyme dose
Improvement of steatorrhea-related complaints | On a weekly base during 9 weeks
  Improvement of complaints (e.g. steatorrhoea, abdominal cramps, abdominal pain).
Change in dietary habits | Week 1, 5 and 9
  Change in dietary habits by means of a food diary
Patient satisfaction | Week 4 and 9
  Patient satisfaction by means of a SF36 questionnaire
Quality of life | week 4 and 9
  Quality of life by means of a SF36 questionnaire
Evaluation of the nutritional status | week 5 and 9
  Evaluation of the nutritional status in the blood and calculating the Body Mass Index (BMI)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Bruno, MD, PhD, Principal Investigator — Department of Gastroeneterology and Hepatology, Erasmus University Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

REFERENCES:
- [Background] Ramo OJ, Puolakkainen PA, Seppala K, Schroder TM. Self-administration of enzyme substitution in the treatment of exocrine pancreatic insufficiency. Scand J Gastroenterol. 1989 Aug;24(6):688-92. doi: 10.3109/00365528909093110. PMID 2479083
- [Background] Czako L, Takacs T, Lonovics J, Lakner L, Dobronte Z, Pronai L, Tulassay Z. [Quality of life in the course of enzyme replacement therapy for chronic pancreatitis]. Orv Hetil. 2002 Jun 23;143(25):1521-7. Hungarian. PMID 12577405
- [Background] Delhaye M, Meuris S, Gohimont AC, Buedts K, Cremer M. Comparative evaluation of a high lipase pancreatic enzyme preparation and a standard pancreatic supplement for treating exocrine pancreatic insufficiency in chronic pancreatitis. Eur J Gastroenterol Hepatol. 1996 Jul;8(7):699-703. PMID 8853261
- [Background] Bruno MJ, Tytgat GN. [4 patients with painless diarrhea and weight loss]. Ned Tijdschr Geneeskd. 1994 Dec 17;138(51):2529-33. No abstract available. Dutch. PMID 7830799